CLINICAL TRIAL: NCT06876142
Title: A Phase 1b/2 Study of Combination Therapy (Mirdametinib and Sirolimus) for RAS Mutated Relapsed Refractory Multiple Myeloma (RRMM)
Brief Title: Combination Therapy (Mirdametinib and Sirolimus) for RAS Mutated Relapsed Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001811; 001811-C
Record Dates: First submitted 2025-03-13; First posted 2025-03-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-07-10

CONDITIONS: Multiple Myeloma; Relapsed and/or Refractory Multiple Myeloma (RRMM)
Keywords: KRAS; NRAS
MeSH Terms: conditions — Multiple Myeloma | interventions — mirdametinib; Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Sirolimus and escalating doses of mirdametinib
  Interventions: Drug: Mirdametinib; Drug: Sirolimus
- Arm 2 (Experimental): Sirolimus and RP2D of mirdametinib
  Interventions: Drug: Mirdametinib; Drug: Sirolimus

INTERVENTIONS:
Drug: Mirdametinib — Capsules taken by mouth twice a day (2-12mg) for days 1-21 days of each 28 day cycle
Drug: Sirolimus — Tablets taken by mouth once a day for days 1-28 days of each 28 day cycle. Loading dose of 12 mg on Day 1 Cycle 1 with 4 mg being taken for the remaining doses.

SUMMARY:
Background:

Multiple myeloma (MM) is a type of blood cancer that affects a person s immunity. MM returns after treatment (relapse) in almost all people; MM may also not respond to initial treatment (refractory). Many people with relapsed refractory MM (RRMM) also have changes in their KRAS and NRAS genes. Researchers want to try a new drug treatment that targets cancer with these changed genes.

Objective:

To test 2 drugs (mirdametinib and sirolimus) in people with RRMM.

Eligibility:

People aged 18 and older with RRMM who have changes in their KRAS or NRAS genes.

Design:

Participants will be screened. They will have blood tests and imaging scans. They will have an eye exam and a test of their heart function. They will need to provide proof of their disease status and of their KRAS or NRAS status. If neither is available, the tests will be repeated.

Participants will have a bone marrow biopsy: A needle will be inserted into a hipbone to draw out some soft tissue.

This study will be done in two parts. In the first part of this study, we will find a safe dose of mirdametinib combined with sirolimus. In the second part, we will learn more about how mirdametinib combined with sirolimus may work against RRMM.

Mirdametinib (capsules) and sirolimus (tablets) are taken by mouth. Participants will take both drugs at home on a 4-week cycle. They will take mirdametinib twice a day for the first 3 weeks of each cycle. They will take sirolimus once a day, every day, during each cycle.

Participants will have study visits once a week during the first cycle, and then on the first day of subsequent cycles. Blood, heart, imaging scans, and other tests will be repeated.

Treatment with the study drugs will go on for 1 year. Then participants will have follow-up visits every 3 months for 4 more years.

DETAILED DESCRIPTION:
Background:

* Multiple myeloma (MM) is the second most prevalent hematologic malignancy. Despite advances in therapy, almost all patients who survive their original presentation eventually relapse. There remains an unmet need in patients who are primary refractory or who have exhausted available therapies.
* To date, the successful therapies in MM have targeted vulnerabilities in myeloma biology such as high protein turnover or overexpressed cell markers. Less success has been had in targeting the molecular pathogenesis or signaling pathways involved in MM oncogenesis.
* RAS mutations can be found in 40-60% of MM tumors and the incidence of RAS mutations goes up with more advanced and heavily pretreated disease.
* The RAS pathway leads to downstream MEK activation which in turn enhances survival, proliferation, and migration of MM cells.
* Preclinical studies suggest that inhibition of both MEK and mTOR is required to impede RAS-dependent pathogenic signaling in MM cells.
* This study will use a MEK inhibitor (mirdametinib) in combination with an mTOR inhibitor (sirolimus) to attempt to block the pathogenic RAS pathway in MM.

Objectives:

* Phase 1b: To determine the recommended phase 2 dose (RP2D) of mirdametinib in combination with sirolimus in participants with RAS mutated relapsed refractory multiple myeloma (RRMM)
* Phase 2: To determine the preliminary efficacy of mirdametinib at RP2D in combination with sirolimus in participants with RAS mutated RRMM as assessed by the overall response rate (ORR) per International Myeloma Working Group (IMWG) criteria

Eligibility:

* Age >= 18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance score <= 2.
* Participants must have a documented diagnosis of MM defined by the International Myeloma Working Group (IMWG) Criteria.
* Participants must have relapsed and/or refractory multiple myeloma (RRMM) with "pentaclass exposed" disease including previous therapy with an anti-CD38 monoclonal antibody, 2 immunomodulatory drugs (IMiDs), and 2 proteasome inhibitors (PIs).
* Participants must have a somatic NRAS or KRAS mutation.

Design:

* This is an open-label, non-randomized, prospective, single-center Phase 1b/2 study evaluating the combination of mirdametinib and sirolimus in participants with RASmutated RRMM.
* During Phase 1b we will find RP2D of mirdametinib in combination with sirolimus using a standard 3 + 3 design.
* During Phase 2 we will use RP2D of mirdametinib in combination with sirolimus to evaluate the efficacy of this combination.
* All participants will receive study drugs for 12 cycles (1 year) or until off-treatment criteria are met. Both drugs will be taken orally daily at home. There will be a one-week break from mirdametinib every cycle (3 weeks on and 1 week off). Sirolimus will be taken continuously.
* Participants will have regular evaluations for safety and response.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have a documented diagnosis of multiple myeloma (MM) defined by the International Myeloma Working Group (IMWG) Criteria. Participants at diagnosis must have had a history of the serum-M protein >= 3 g/dL and or bone marrow plasma cells >= 10% and the history of at least one of the following:

  * Anemia: hemoglobin <= 10 g/dL or a 2g/dL decrease from the lower limit of normal,

OR

* Renal failure: creatinine clearance < 40 ml/min, OR
* Hypercalcemia: calcium (Ca) >= 11 mg/dL OR > 1 mg/dL higher than the upper limit of normal (ULN), OR
* Lytic bone lesions on X-Ray, Computed Tomography (CT), or Positron Emission Tomography (PET)/CT, OR
* >= 2 focal lesions on spinal Magnetic Resonance Imaging (MRI), OR
* >= 60% bone marrow plasma cells, OR
* Involved/un-involved serum-free light chain ratio >= 100.

  * Participants must have measurable disease per International Myeloma Working Group (IMWG) criteria.
  * Participants must have relapsed and/or refractory multiple myeloma (RRMM) with "penta-class exposed" disease, as defined by previous therapy with an anti-CD38 monoclonal antibody, 2 immunomodulatory drugs [IMiDs], and 2 proteasome inhibitors [Pis]), 3 previous lines of therapy, and no other available options.
  * Participants must have a history of known somatic mutation in KRAS or NRAS. Note: For participants that come to NIH without confirmation of KRAS or NRAS, their status will be determined by the TSO500 NSR device.
  * Participants must be off other myeloma-directed therapy (except for radiation) for at least 14 days prior to the study treatment initiation.
  * Age >= 18 years.
  * ECOG performance status <= 2.
  * Participants must have adequate organ and marrow function as defined below:

Absolute neutrophil count (ANC): >= 1,000 cells/microliter

Platelets: >= 75,000 cells/microliter

Total bilirubin: within normal institutional limits

Aspartate Aminotransferase (AST): <= 3 X ULN

Alanine Aminotransferase (ALT): <= 3 X ULN

Renal function: creatinine clearance (CrCl) >= 40 mL/min calculated by Cockcroft-Gault,

-Individuals of childbearing potential (IOCBP) must agree to use highly effective contraception (hormonal, intrauterine device [IUD], abstinence, surgical sterilization) at the study entry and for at least 12 weeks after the last dose of sirolimus or 6 months after the last dose of mirdametinib, whichever is longer. Barrier methods such as condoms (male or female) or occlusive caps (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream or vaginal suppository must be used in addition to hormonal contraception. Note: IOCBP is defined as any individual who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal.

Individuals able to father a child must agree to use an effective method of contraception (barrier plus spermicide, surgical sterilization, abstinence) at the study entry and for 3 months after the last dose of mirdametinib. We also will recommend individuals able to father a child with partners of childbearing potential ask partners to be on highly effective birth control (hormonal, IUD, surgical sterilization) for at least 3 months after the last dose of mirdametinib. Individuals able to father a child must not freeze or donate sperm within the same period.

* Breastfeeding participants must be willing to discontinue breastfeeding after study treatment initiation.
* Participants seropositive for human immunodeficiency virus (HIV) infection must:

  * be on anti-retroviral therapy; and
  * have the undetectable viral load.
* Participants seropositive for Hepatitis C virus (HCV) infection must

  * have been treated and cured; or
  * if currently on treatment, have an undetectable HCV viral load.
* Participants seropositive for Hepatitis B virus (HBV) infection must
* be on suppressive therapy if necessary; and
* have viral load <100 IU/mL.
* Ability of the participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Received any investigational agents within 14 days prior to the study treatment initiation.
* Vaccinated with live, attenuated vaccines within 30 days prior to the study treatment initiation.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to mirdametinib and/or sirolimus.
* Current diagnosis of plasma cell leukemia.
* Current or history of amyloidosis.
* Current or history of New York Heart Association (NYHA) Stage III or IV heart failure
* Current or history of Interstitial Lung Disease.
* Current or history of glaucoma and/or an intraocular pressure > 22 mmHg, retinal pigment epithelial detachment, or other primary ocular/retinal diseases.
* Current or history of retinal vein occlusion (RVO).
* Comorbidities that put undue risk of RVO such as uncontrolled hypertension (chronic systolic blood pressures > 160 mm Hg) and/or uncontrolled diabetes mellitus type II (DMII) (chronic clinical signs/symptoms of hyperglycemia; diabetic participants must have a hemoglobin A1c value < 9% to be eligible).
* Participants receiving systemic or ocular glucocorticoid therapy equivalent to > 10 mg of prednisone daily within 14 days prior to the study treatment initiation. Note: Participants with endocrine deficiencies, who receive physiologic, or stress doses of steroids are eligible.
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 within 14 days prior to the study treatment initiation. Lists including medications and substances known or with the potential to interact with the CYP3A4 isoenzymes are provided here: http://medicine.iupui.edu/clinpharm/ddis/table.aspx.
* Participants receiving any medications or substances that are strong inhibitors of breast cancer resistance protein (BCRP) within 14 days prior to the study treatment initiation (i.e., curcumin, cyclosporine, darolutamide, eltrombopag, febuxostat, fostamatinib, rolapitant, sofosbuvir and velpatasvir and voxilaprevir, and teriflunomide).
* Positive beta-human chorionic gonadotropin (beta-HCG) serum or urine pregnancy test performed in IOCBP at screening.
* Participant has abnormal QT interval corrected by Fridericia s formula (QTcF >470 ms, as determined by the mean QTcF values from the ECG assessments at screening (one triplicate).
* Uncontrolled intercurrent illness or factors evaluated by medical history and physical exam that would potentially increase the risk of the participant.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2033-01-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: determine the RP2D of the mirdametinib in combination with sirolimus in participants with RAS-mutated RRMM | 28 days
  The RP2D will be determined by the dose found in the 3+3 design to cause < 33% toxicity as defined by the DLT criteria.
Phase 2: determine the preliminary efficacy of mirdametinib at RP2D in combination with sirolimus in participants with RAS-mutated RRMM as assessed by the ORR per IMWG | Day 1 of every cycle, at suspected CR, End of cycles 6 and 12, Safety Follow Up visit, every 3 months after that until progression, initiation of another line of therapy, or 5 years since treatment initiation.
  The fraction of participants with a RAS mutation who experience a response (PR, VGPR, CR, or sCR) while on the study treatment will be determined by dividing the number of responders by the total number of evaluable participants. The fraction will be reported along 95% two-sided confidence intervals.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Day 1 of every cycle, at suspected CR, End of cycles 6 and 12, Safety Follow Up visit, every 3 months after that until progression, initiation of another line of therapy, or 5 years since treatment initiation.
  DOR will be assess with blood tests and radiographic findings and reported using the Kaplan-Meier method.
Progression Free Survival (PFS) | Day 1 of every cycle, at suspected CR, End of cycles 6 and 12, Safety Follow Up visit, every 3 months after that until progression, initiation of another line of therapy, or 5 years since treatment initiation.
  PFS will be assessed with blood tests and radiographic findings and reported using the Kaplan-Meier method.
Overall Survival (OS) | Day 1 of every cycle, EOT, Safety Follow-up visit, then every 3 months(+/-2 weeks) until disease progression or the initiation of another line of therapy for up to 5 years after the treatment initiation. After progression or initiation of a new treatment
  OS will be assessed and reported using the Kaplan-Meier method and include any cause of death.
Safety | Until 30 days after the last dose of study agents
  The number and frequency of adverse events for participants as assessed per CTCAE version 5. Safety will be analyzed by reporting the number of patients experiencing toxicity, classified by type and grade to the experimental regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Hill, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be made available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available upon request and with the permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001811-C.html